CLINICAL TRIAL: NCT02232347
Title: Effect of Ketamine Versus Sufentanil on Cerebral Glutamate After Traumatic Brain Injury : a Randomized, Double-blinded, Microdialysis Study
Brief Title: Ketamine and Glutamate After Brain Injury : a Microdialysis Study
Acronym: KETABRAIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pierre-Julien CUNGI (Other)
Responsible Party: Sponsor-Investigator, Pierre-Julien CUNGI, MD, Direction Centrale du Service de Santé des Armées
Organization: Direction Centrale du Service de Santé des Armées (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCSSA KETABRAIN
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Head Trauma
Keywords: traumatic brain injury; ketamine; microdialysis; PtiO2; glutamate
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic | interventions — Ketamine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine (Experimental): ketamine 5 mg/kg/h, continuous infusion for 48 hours
  Interventions: Drug: Ketamine
- sufentanil (Active Comparator): sufentanil 0,5 mcg/kg/h, continuous infusion for 48 hours
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Ketamine
  Arms: ketamine
Drug: Sufentanil
  Arms: sufentanil

SUMMARY:
The objective of the study is to compare the effects of 48 hours ketamine infusion versus sufentanil infusion on brain glutamate concentrations measured with microdialysis after traumatic brain injury.

We hypothesize that ketamine infusion will decrease high glutamate values faster than sufentanil.

DETAILED DESCRIPTION:
Inclusion of 20 consecutive head trauma patients. Randomization and double-blind to compare the effects of ketamine versus sufentanil on brain glutamate concentrations measured with microdialysis.

Ketamine is an anti-N-methyl-D-aspartate (NMDA) medication. It is supposed to limit excitotoxicity of amino-acids, especially glutamate. Glutamate is known to be elevated in more than 60% of the severe head trauma patients. It induces cortical spreading depression which can aggravate prognosis. It's a daily used medication in anesthesia and intensive care units for sedation and induction of anesthesia. It's the recommended medication for induction of unstable wounded soldiers on the field because of its neutrality on haemodynamic state.

Sufentanil is the reference opioid for sedation in ICU in Europe. It can induce hypotension which is deleterious for cerebral perfusion pressure after brain trauma.

In our unit, patients with severe head injury are monitored by a triple lumen access device including ICP (IntraCerebral Pressure), PtiO2 (oxygen pressure in the brain) and microdialysis. This last monitoring allows measurement of brain parenchymal concentrations of small molecules : glucose, lactate, pyruvate, glutamate, glycerol,.... It's a tool to evaluate the metabolic state of the brain divided into 4 categories : normal, hyperglycolysis, ischemia and metabolic crisis.

Then, we will detail the effects of ketamine on metabolic state of the brain, especially glutamate concentration. Normal values are below 10 micromol/ml. After head trauma it can dramatically increase to values up to 50 or even 100 micromol/ml, with normalization after 24 hours. Ketamine is expected to decrease these high values faster than described in observational studies.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Glasgow Coma Scale (GCS) < 9
* > 3 days of sedation expected at the arrival

Exclusion Criteria:

* pregnancy
* < 18 years old
* estimated survival < 48 hours post-trauma
* expected sedation < 3 days
* coagulation impairment (platelets<100.000/mm3 and prothrombin time (TP) <60%)
* Cardiac arrest before ICU admission
* Admission > 12 hours after trauma
* Multimodal monitoring implanted > 24 hours post trauma
* Participation to the study refused by the next of kind
* No next of kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
brain glutamate concentrations | H0-H12, H12-H24, H24-H36 and H36-H48
  To compare the kinetic of brain glutamate concentration decrease during 4 periods of 12 hours between ketamine infusion group (KET) and sufentanil standard infusion group (STD)

SECONDARY OUTCOMES:
metabolic profile | H0-H12, H12-H24, H24-H36 and H36-H48
  To compare the brain metabolic profile (normal, ischemic, hyperglycolytic and metabolic crisis) of the patients related to their group of treatment : ketamine (KET) and sufentanil (STD) by measuring brain glucose, brain lactate, brain glycerol concentrations and brain lactate/pyruvate ratio.
Episodes of intracranial hypertension (ICHT) and brain ischemia | H0-H12, H12-H24, H24-H36 and H36-H48
  To compare the number of ICHT episodes (ICP>20 mm Hg more than 15 minutes) and to compare the number of ischemic episodes (PtiO2<20 mm Hg more than 15 minutes) between the 2 groups
Therapeutic Intensity Level (TIL) | Days 1 and 2
  To compare the TIL value between the 2 groups. TIL is a score developed to measure the intensity of cares for head trauma patients. Lower scores are meaning less intense cares. It is calculated for 24 hours periods.
Glasgow Outcome Scale (GOS) et extended Glasgow Outcome Scale (eGOS) | 6 months and 1 year
  To describe the prognosis of the patients of the KETAMINE group versus SUFENTANIL group. GOS is the international validated score for evaluation of the prognosis after head trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Ambroise MONTCRIOL, MD, Principal Investigator — Direction Centrale du Service de Santé des Armées
Locations (1):
- Sainte Anne Military Teaching Hospital, Toulon, France

REFERENCES:
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. I. Blood pressure and oxygenation. J Neurotrauma. 2007;24 Suppl 1:S7-13. doi: 10.1089/neu.2007.9995. No abstract available. PMID 17511549
- [Background] Hughes S. Towards evidence based emergency medicine: best BETs from the Manchester Royal Infirmary. BET 3: is ketamine a viable induction agent for the trauma patient with potential brain injury. Emerg Med J. 2011 Dec;28(12):1076-7. doi: 10.1136/emermed-2011-200891. PMID 22101599
- [Background] Filanovsky Y, Miller P, Kao J. Myth: Ketamine should not be used as an induction agent for intubation in patients with head injury. CJEM. 2010 Mar;12(2):154-7. doi: 10.1017/s1481803500012197. No abstract available. PMID 20219164
- [Background] Hudetz JA, Pagel PS. Neuroprotection by ketamine: a review of the experimental and clinical evidence. J Cardiothorac Vasc Anesth. 2010 Feb;24(1):131-42. doi: 10.1053/j.jvca.2009.05.008. Epub 2009 Jul 29. No abstract available. PMID 19640746
- [Background] Ward JL, Harting MT, Cox CS Jr, Mercer DW. Effects of ketamine on endotoxin and traumatic brain injury induced cytokine production in the rat. J Trauma. 2011 Jun;70(6):1471-9. doi: 10.1097/TA.0b013e31821c38bd. PMID 21817985
- [Background] Bhutta AT, Schmitz ML, Swearingen C, James LP, Wardbegnoche WL, Lindquist DM, Glasier CM, Tuzcu V, Prodhan P, Dyamenahalli U, Imamura M, Jaquiss RD, Anand KJ. Ketamine as a neuroprotective and anti-inflammatory agent in children undergoing surgery on cardiopulmonary bypass: a pilot randomized, double-blind, placebo-controlled trial. Pediatr Crit Care Med. 2012 May;13(3):328-37. doi: 10.1097/PCC.0b013e31822f18f9. PMID 21926656
- [Background] Sakowitz OW, Kiening KL, Krajewski KL, Sarrafzadeh AS, Fabricius M, Strong AJ, Unterberg AW, Dreier JP. Preliminary evidence that ketamine inhibits spreading depolarizations in acute human brain injury. Stroke. 2009 Aug;40(8):e519-22. doi: 10.1161/STROKEAHA.109.549303. Epub 2009 Jun 11. PMID 19520992
- [Background] Hartings JA, Bullock MR, Okonkwo DO, Murray LS, Murray GD, Fabricius M, Maas AI, Woitzik J, Sakowitz O, Mathern B, Roozenbeek B, Lingsma H, Dreier JP, Puccio AM, Shutter LA, Pahl C, Strong AJ; Co-Operative Study on Brain Injury Depolarisations. Spreading depolarisations and outcome after traumatic brain injury: a prospective observational study. Lancet Neurol. 2011 Dec;10(12):1058-64. doi: 10.1016/S1474-4422(11)70243-5. Epub 2011 Nov 3. PMID 22056157
- [Background] Raboel PH, Bartek J Jr, Andresen M, Bellander BM, Romner B. Intracranial Pressure Monitoring: Invasive versus Non-Invasive Methods-A Review. Crit Care Res Pract. 2012;2012:950393. doi: 10.1155/2012/950393. Epub 2012 Jun 8. PMID 22720148
- [Background] Stuart RM, Schmidt M, Kurtz P, Waziri A, Helbok R, Mayer SA, Lee K, Badjatia N, Hirsch LJ, Connolly ES, Claassen J. Intracranial multimodal monitoring for acute brain injury: a single institution review of current practices. Neurocrit Care. 2010 Apr;12(2):188-98. doi: 10.1007/s12028-010-9330-9. PMID 20107926
- [Background] Bourgoin A, Albanese J, Wereszczynski N, Charbit M, Vialet R, Martin C. Safety of sedation with ketamine in severe head injury patients: comparison with sufentanil. Crit Care Med. 2003 Mar;31(3):711-7. doi: 10.1097/01.CCM.0000044505.24727.16. PMID 12626974
- [Background] Bourgoin A, Albanese J, Leone M, Sampol-Manos E, Viviand X, Martin C. Effects of sufentanil or ketamine administered in target-controlled infusion on the cerebral hemodynamics of severely brain-injured patients. Crit Care Med. 2005 May;33(5):1109-13. doi: 10.1097/01.ccm.0000162491.26292.98. PMID 15891344
- [Background] Chamoun R, Suki D, Gopinath SP, Goodman JC, Robertson C. Role of extracellular glutamate measured by cerebral microdialysis in severe traumatic brain injury. J Neurosurg. 2010 Sep;113(3):564-70. doi: 10.3171/2009.12.JNS09689. PMID 20113156